CLINICAL TRIAL: NCT05523661
Title: The Safety and Clinical Efficacy of Dasatinib Plus Human CD19/CD22 Bispecific CAR-T Cell Therapy for Elderly Subjects With Ph-positive Acute Lymphoblastic Leukemia
Brief Title: Dasatinib Plus Anti-CD19/CD22 Bispecific CAR-T Cell Therapy for Elderly Ph-positive ALL Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, principal investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-ALL02-POC
Record Dates: First submitted 2021-11-14; First posted 2022-08-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Ph Positive ALL; CAR-T Cell; Dasatinib
Keywords: CD19/CD22 Bispecific CAR-T; Ph-positive lymphoblastic leukemia; Dasatinib
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib plus anti-CD19/CD22 CAR-T cells (Experimental): Administration with oral Dasatinib plus anti-CD19/ CD22 CAR-T cells in the elderly Ph-positive ALL patients.
  Interventions: Drug: Dasatinib plus anti-CD19/CD22 CAR-T cells

INTERVENTIONS:
Drug: Dasatinib plus anti-CD19/CD22 CAR-T cells — Dasatinib plus VP chemotherapy was administrated to newly diagnosed Ph-positive patients aged 55-70 years old,if hCR was achieved,autolymphocyte was collected,and anti-CD19/CD22 CAR-T cells infusion was administrated to patients followed by Fludarabine and Cyclophosphamide therapy

SUMMARY:
To evaluate the safety and efficacy of Dasatinib plus CD19/CD22 Bispecific CAR-T for the treatment of elderly Ph-positive lymphoblastic leukemia. Newly diagnosed Ph-positive patients will be given Dasatinib plus VP chemotherapy for induction treatment,if a hematologic complete remission was observed then a lymphocyte collection will be administrated to patients. Then chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19/CD22 CAR+ T cells

DETAILED DESCRIPTION:
Newly diagnosed ph-positive ALL patients over 60 and less than 70 years old will be enrolled. Patients will be given Dasatinib plus VP chemotherapy for induction remission treatment, if a hematologic complete remission was observed then a lymphocyte collection will be administrated to patients. Then chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19/CD22 CAR+ T cells

ELIGIBILITY:
Inclusion Criteria:

* (1)55 to 70 Years Old, Male and female;
* (2) Newly diagnosed Ph-positive ALL
* (3) ECOG score 0-1;
* (4) The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators;
* (5) Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Creatinine is in the normal range;
  2. Left ventricular ejection fraction >50%;
  3. Baseline oxygen saturation>92%;
  4. Total bilirubin ≤ 1.5×ULN;
  5. ALT and AST ≤ 2.5×ULN;
* (6) Able to understand and sign the Informed Consent Document

Exclusion Criteria:

* (1) Disease relapse;
* (2) Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
* （3) ECOG >=2 during CAR-T therapy
* (4) Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease; Heart disease including the following condition

  1. Ultrasound shows left ventricular ejection fraction <50%;
  2. stable/unstable angina,myocardia infarction
  3. Baseline oxygen saturation>92%;
  4. history of pacemaker inplantation
  5. more than 2 leads ST segments decrease>1mm,or more than 2 consecutive leads T wave inversion;
  6. Long QT syndrom
  7. A severe arrhythmia requiring medical treatments
  8. bradycardia,HR<50BPM I.QTc>450ms
* (5)Uncontrolled infection during screening peroid; Hemodynamic instability associated with infection,a new infection or aggravation of the original infection;new lesions on imaging;fever of unkown cause
* (6) Patients with symptoms of central nervous system;greater than grade 2 requring treatment,paralysis,aphasia,acute cerebral infarction,severe traumatic brain injury,schizophrenia
* (7)Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
* (8) HIV infection
* (9)Subjects with positive HBsAg or HBcAb and peripheral blood HBV DNA titer detection ≥ 1 × 102 copy number / L; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; CMV DNA positive; syphilis positive;
* (10) Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* (11) allergy to Dasatinib
* (12) history of autoimmune disaese

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving molecular CR | 3 months after infusion of Anti-CD19/CD22 CAR-T cells
  number of patients achieving molecular CR

SECONDARY OUTCOMES:
OS for patients receiving infusion of anti-CD19/CD22 CAR-T cells | 2-year OS
  Overall survival for all patients enrolled
RFS for patients receiving infusion of anti-CD19/CD22 CAR-T cells | 2-year RFS
  Relapse free survival for all patients enrolled
Number of patients achieving molecular CR | 6 months after infusion of Anti-CD19/CD22 CAR-T cells
  number of patients achieving molecular CR after infusion of Anti-CD19/CD22 CAR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moorman AV, Harrison CJ, Buck GA, Richards SM, Secker-Walker LM, Martineau M, Vance GH, Cherry AM, Higgins RR, Fielding AK, Foroni L, Paietta E, Tallman MS, Litzow MR, Wiernik PH, Rowe JM, Goldstone AH, Dewald GW; Adult Leukaemia Working Party, Medical Research Council/National Cancer Research Institute. Karyotype is an independent prognostic factor in adult acute lymphoblastic leukemia (ALL): analysis of cytogenetic data from patients treated on the Medical Research Council (MRC) UKALLXII/Eastern Cooperative Oncology Group (ECOG) 2993 trial. Blood. 2007 Apr 15;109(8):3189-97. doi: 10.1182/blood-2006-10-051912. Epub 2006 Dec 14. PMID 17170120
- [Background] Short NJ, Kantarjian H, Jabbour E, Ravandi F. Novel Therapies for Older Adults With Acute Lymphoblastic Leukemia. Curr Hematol Malig Rep. 2018 Apr;13(2):91-99. doi: 10.1007/s11899-018-0440-3. PMID 29423571